CLINICAL TRIAL: NCT02847416
Title: to Explore the Characteristics of Mean Airway Pressure, Oscillatory Amplitude and Power Spectral Density (PSD) of Oscillatory Airway Pressure That Generate by Various Loaded and Flow Rate During Expiration and Inspiration in Healthy Subjects
Brief Title: A Study of Pressure and Flow Characteristics During Inspiration and Expiration Using BreatheMAX® in Healthy Subjects
Acronym: PFBM
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Khon Kaen University (Other)
Responsible Party: Principal Investigator, Sujittra Kluayhomthong, Principle Inveatigator, Khon Kaen University
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Other
Other Study IDs: KKU2016
Record Dates: First submitted 2016-07-25; First posted 2016-07-28 (Estimated); Last update posted 2018-03-05 (Actual); Status verified 2017-08

CONDITIONS: Healthy Subjects

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Inspiratory group (Experimental): the subjects will be instructed to inspire as deeply as possible with steady flow rate for 3 seconds with end-inspiratory pause for 2-3 seconds through the inspiratory circuit and follow by passive exhalation
  Interventions: Device: BreatheMAX breathing device
- expiratory group (Experimental): the subjects will be instructed to inspire as deeply as possible through the nose with end-inspiratory pause for 2-3 seconds and partially forced exhalation with reach to 1/3 of expiratory reserve volume (ERV) for at least 3 seconds through expiratory circuit
  Interventions: Device: BreatheMAX breathing device

INTERVENTIONS:
Device: BreatheMAX breathing device

SUMMARY:
the aim of this study are to explore the characteristics of mean airway pressure, oscillatory amplitude and power spectral density (PSD) of oscillatory airway pressure that generate by various loaded and flow rate during expiration and inspiration in healthy subjects and to explore the best loaded and flow rate for airway secretion clearance using the BreatheMAX® device

DETAILED DESCRIPTION:
For inspiratory group, the resistive load 3, 4, 5, 6 and 7 cm H2O were test with three flow rate: 0.2, 0.4, and 0.6 L/sec in each load. In each flow rate, the subjects were instructed to inspire as deeply as possible with steady flow rate for 3 seconds with end-inspiratory pause for 2-3 seconds through the inspiratory circuit and follow by passive exhalation. For expiratory group, the resistive load and flow rate were test similar inspiratory group. In each flow rate, the subjects were instructed to inspire as deeply as possible through the nose with end-inspiratory pause for 2-3 seconds and partially forced exhalation with reach to 1/3 of expiratory reserve volume (ERV) for at least 3 seconds through expiratory circuit

ELIGIBILITY:
Inclusion Criteria:

* the healthy subjects
* able to breathe against resistive load with the BreatheMAX device
* good conscious and cooperation

Exclusion Criteria:

- fever

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 10 (Actual)
Dates: Start 2016-08; Primary Completion 2017-07 (Actual); Study Completion 2017-08-28 (Actual)

PRIMARY OUTCOMES:
PSD of oscillatory airway pressure | 5 seconds during inspiration and expiration testing period

SECONDARY OUTCOMES:
mean airway pressure | 5 seconds during inspiration and expiration testing period
oscillatory amplitude | 5 seconds during inspiration and expiration testing period

CONTACTS AND LOCATIONS:
Overall Officials: sujittra Kluayhomthong, master degree, Principal Investigator — faculty of associated medical science, KhonKaen University, Thailand 40002
Locations (1):
- Pulmonary research room of physical therapy department, Faculty of associated medical sciences, Khon Kaen University, Khon Kaen, Thailand

IPD SHARING:
Plan to Share IPD: Undecided